CLINICAL TRIAL: NCT04947397
Title: Investigation of Pupillometry as Guide for Extubation Readiness in Anesthetized Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-32664
Record Dates: First submitted 2021-06-11; First posted 2021-07-01 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Anesthesia; Laryngospasm on Emergence
Keywords: Pediatric; Anesthesia; Extubation; Pupillometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 (No Intervention): Traditional deep extubation at 1.5 minimum alveolar concentration (MAC)
- Group 2 (Experimental): Deep extubation guided by pupillometry -- at < 0.5 MAC of vapor + propofol and fentanyl
  Interventions: Diagnostic Test: Pupillometry

INTERVENTIONS:
Diagnostic Test: Pupillometry — Pupillometry prior to extubation
  Arms: Group 2

SUMMARY:
Investigation of pupillometry as guide for extubation readiness in anesthetized children.

DETAILED DESCRIPTION:
Can a pupil metric be used to make extubation more safe in anesthetized children?

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing general anesthesia and endotracheal intubation for surgery.
* American Society of Anesthesiologists Physical Status Class I and II patients.

Exclusion Criteria:

* Central nervous system abnormality.
* Ophthalmologic abnormality.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Abelson, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- UCSF Benioff Children's Hospital Oakland, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] — Age range: 2 years old through 10 years old
  years | 4.4 (2.9) | 5.5 (3.2) | 5.0 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Not collected because not relevant. Pupillometry is not considered dependent on whether male or female.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Extubation Success
Description: Maintenance of spontaneous ventilation without pathologic airway response such as laryngospasm.
  Ventilation monitored in a standard manner, using chest wall movement, capnography, reservoir bag movement, condensation of anesthetic mask and auscultation.
Time Frame: Immediately after extubation
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 10
Participants | 10 | 10

2. Secondary Outcome: Anesthetic Vapor Concentration at Extubation
Description: Percent of end-tidal sevoflurane at extubation
Time Frame: At the time of extubation
Measure: Mean (Standard Deviation); unit: Percent of sevoflurane
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 10
Percent of sevoflurane | 3.8 (0) | 0.8 (0.1)

3. Other Pre Specified Outcome: Breath-holding
Description: Measurement tool: Capnogram
Time Frame: Prior to extubation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data were collected over the time period spanning extubation to discharge from the PACU, a time range of 1 to 3 hours.
Description: Extubation of the trachea in pediatric anesthesia has inherent risks. Risks include airway compromise secondary to laryngospasm, bronchospasm or other forms of airway obstruction.
  When severe, airway compromise can lead to cardiac arrest.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT04947397/Prot_SAP_003.pdf